CLINICAL TRIAL: NCT06506188
Title: UNCPM 22402 - Leveraging Infant Visit PrEP INtegration & tasK Shifting to Improve Post-partum HIV Prevention in Malawi
Brief Title: Leveraging Infant Visit PrEP INtegration & tasK Shifting to Improve Post-partum HIV Prevention in Malawi
Acronym: LINK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0323; 1P01HD112215 (NIH)
Record Dates: First submitted 2024-06-26; First posted 2024-07-17 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Breastfeeding; HIV Prevention
Keywords: Breastfeeding; HIV
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: This is an effectiveness-implementation type I hybrid cluster randomized trial which includes prospective data collection (both quantitative and qualitative) as well as use of existing surveillance data to inform pre-defined effectiveness and implementation outcomes of interest. Randomization and implementation of the LINK model occurs at the clinic level, and individuals are considered exposed or unexposed based on their attendance at intervention or control clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LINK model (Experimental): Women at these sites receive the LINK model, which includes integrated EPI/HIV testing, screening for HIV risk, support for male partner engagement, and community-facility linkage (CFL) peer moms for breastfeeding women using PrEP for ongoing support and follow-up for breastfeeding women who disengage from PrEP care. This model is integrated into the SOC and does not replace SOC activities.
  Interventions: Behavioral: LINK model
- Standard of Care (No Intervention): Women at these sites continue to receive the current standard of care (SOC) for postpartum HIV testing, PrEP screening, and PrEP care in Malawi.

INTERVENTIONS:
Behavioral: LINK model — The LINK model includes four elements:
  (1) linking postpartum HIV testing and PrEP services to early infant vaccination, (2) screening for HIV risk among those who test negative for HIV at the early infant vaccination visit, (3) male partner engagement to support status awareness within couples and PrEP persistence, and (4) community-facility linkage (CFL) peer mom for ongoing support of breastfeeding women using PrEP and follow-up of breastfeeding women who disengage from PrEP care.
  Arms: LINK model

SUMMARY:
The goal of the Leveraging Infant Visit PrEP INtegration & tasK Shifting to Improve Postpartum HIV Prevention in Malawi (LINK) study is to evaluate both the effectiveness of a postpartum prevention package ("LINK model") among post-partum women and its implementation into existing clinical care models in Lilongwe, Malawi. The main question the study seeks to answer is:

Do women at clinics implementing the LINK model have improved Pre-exposure Prophylaxis (PrEP) persistence compared to women at clinics receiving the standard of care?

Researchers will compare the LINK model to standard of care by randomizing twelve sites to either the LINK model or the standard of care. Then researchers will review existing medical record and health surveillance data, and qualitative and quantitative data collected from intervention and control sites.

DETAILED DESCRIPTION:
Study Design Overview:

The LINK study is an effectiveness-implementation type I hybrid cluster randomized trial. Prospective data collection and existing medical record and health surveillance data will be used to evaluate the effectiveness and implementation of the LINK model. The LINK model is a clinical intervention aiming to improve PrEP persistence among postpartum women. Outcomes from this trial will be used to assess its potential for implementation outside of the trial setting.

The study will take place in Lilongwe district in Malawi, a priority district for HIV prevention services given high HIV incidence. Twelve sites in Lilongwe will be randomized 1:1 to the LINK model or the standard of care.

The LINK model includes:

1. Linking postpartum HIV testing and PrEP services to early infant vaccination
2. Screening for HIV risk among those who test negative for HIV at the early infant vaccination visit
3. Male partner engagement to support status awareness within couples and PrEP persistence
4. Community facility-linkage (CFL) peer mom for ongoing support of breastfeeding moms using PrEP, and follow-up of breastfeeding women who disengage from PrEP care

Components #1-3 are directly integrated into the Expanded Programme on Immunization (EPI) infant vaccination visit and will be carried out by a mix of existing staff and study-hired HIV diagnostic assistants (HDA). HDAs are a lower healthcare worker cadre that Malawi has successfully deployed to expand HIV testing services. Component #4 will take place outside of the infant immunization clinic, integrated into existing PrEP clinics and clinic flow at each site. Component #4 will shift the tasks of engaging women, exploring strategies to facilitate ongoing PrEP care attendance, and tracing persons who disengage from care from the the PrEP prescriber (typically a nurse) to the CFL "PrEP peer" mother. The study anticipates supporting placement of one PrEP-trained HDA and at least one CFL "PrEP peer" at each intervention site. All PrEP services, including clinical evaluation and medication refill or administration, will be provided by Malawi Ministry of Health (MoH) and/or local implementing partners tasked with PrEP delivery.

Data collection methods will include structured observation, medical record review, surveys, and in-depth interviews (IDI) with patients in each of the twelve clinics. The primary outcome, PrEP persistence, will be assessed by PrEP medical record review of patients at intervention and control clinics. Additionally, there will be study-specific data collection tools including surveys, IDI, and dried blood spots (DBS) administered to participants consented and enrolled into the study at intervention and control clinics. Participants will not be followed longitudinally. Study data assistants will administer surveys at each participating site for women receiving services related to infant vaccines and PrEP care. These surveys will collect demographic information, HIV risks, and PrEP utilization (if applicable). Researchers will collect DBS from a subset of women who initiated PrEP to measure oral PrEP adherence.

A subset of women in intervention clinics, including those receiving services at the PrEP and/or EPI clinics, as well as clinical providers, implementing partners, and members of the Malawi Ministry of Health will be asked to participate in an IDI focused on acceptability and feasibility of the intervention. For women, interviews will focus on experiences with each component of the intervention and partner support for HIV testing and PrEP usage during the postpartum period. Non-patient stakeholders' interviews will focus on context and feasibility of implementation, scale, and sustainability of the LINK model.

ELIGIBILITY:
PrEP user cohort:

PrEP user cohort includes all adolescent and adult women >=15 years old who are on PrEP and breastfeeding, enrolled in PrEP at each of the participating 12 sites during the study follow-up period. PrEP provision and clinical management will be at the discretion of the non-study PrEP providers according to Malawi PrEP guidelines and eligibility. Data for these women are abstracted from PrEP records. We are seeking a waiver of informed consent for all health record abstraction for the LINK study.

Inclusion criteria:

* Female enrolled in PrEP care at a study site
* Breastfeeding documented while on PrEP
* Living without HIV

Exclusion criteria:

- None

PrEP user survey and dried blood spot sub-group Breastfeeding women 15 years and older who are presenting ~6 months after initiating PrEP are eligible participation in study surveys and dried blood spot using fingerstick specimen collection. Women aged 15-17 will be asked to provide assent with parental/guardian consent. Every woman who is consented for the survey will also be asked about their willingness to participate in in-depth interviews. Only a subset of consenting participants, purposively sampled to reflect variety in key demographics and clinical metrics, will complete interviews.

Inclusion criteria:

* Female who has presented for PrEP visit at a participating clinical site at least ~6 months after initiating PrEP
* Aged 15 years (assent with parental/guardian consent for women aged 15-17)
* Living without HIV

Exclusion criteria:

- Decline informed consent

Postpartum women - health passport review We review use existing health records (Health passports) of postpartum women presenting to infant immunization appointments with their child. No identifying information will be collected from this group.

Inclusion criteria:

- Female presenting with infant under 3 for under-five visit to participating clinical site

Exclusion criteria:

- None

Postpartum women - surveys Postpartum women 15 years and older who are presenting to under-five visits with their child under 3 will be eligible for participation in study surveys. Women aged 15-17 will be asked to provide assent with parental/guardian consent. Every woman who is consented for the survey will also be asked about their willingness to participate in in-depth interviews. Only a subset of consenting participants, purposively sampled to reflect variety in key demographics and clinical metrics, will complete interviews.

Inclusion criteria:

* Female presenting for child vaccination to participating clinical site
* Aged15 years and older (assent with parental/guardian consent for women aged 15-17)

Exclusion criteria:

- Decline informed consent

Non-patient key stakeholder Non-patient stakeholders relevant to intervention implementation at the clinic and national level, including clinical and policy stakeholders. Examples of clinical stakeholders may include key clinic staff working in PrEP, HIV testing, EPI, and CFL peer support mothers. Policy and implementing partner stakeholders may include officials from the Malawi Ministry of Health, donors in HIV prevention (e.g. PEPFAR, the Global Fund), members of community advocacy groups, the Lilongwe DHO, and other persons involved in infant vaccine and HIV prevention program and policy development and implementation in HIV prevention in Lilongwe.

Inclusion criteria:

* Aged 18 years and older
* Involved in relevant activities pertinent to integration or provision of PrEP services such as PrEP providers, peer mothers, HIV diagnostic assistants, or clinic managers, OR policy and implementing partner stakeholders such as officials from the Malawi Ministry of Health, donors in HIV prevention (e.g. PEPFAR, the Global Fund), members of community advocacy groups, the Lilongwe DHO, and other persons involved in infant vaccine and HIV prevention program and policy development and implementation in HIV prevention in Lilongwe

Exclusion criteria:

- Decline informed consent

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
PrEP persistence: Proportion of patients on PrEP for 6 months after initiation with no lapse of PrEP coverage exceeding 14 days | PrEP initiation or initiation of breastfeeding while on PrEP through 6 months
  Proportion of breastfeeding patients with health record-reported PrEP use (oral or injectable) who maintain ongoing PrEP usage with no more than a 14-day lapse of expected available pills or timely injections from oral or injectable PrEP approximately 6 months after PrEP initiation, among the total number of breastfeeding patients with health record-reported PrEP use (oral or injectable)
PrEP uptake: Proportion of patients initiating PrEP while breastfeeding among HIV-negative deliveries at the clinic in the past year | Study start to study end (approximately 3.5 years)
  Proportion of number of breastfeeding patients with record-reported initiation of PrEP (oral or injectable) in the study period, among HIV-negative deliveries in a clinic in the study period
Oral PrEP adherence: Proportion of patients on oral PrEP with PrEP metabolite levels consistent with >=4 pills per week at a 6-month oral PrEP visit | PrEP initiation or initiation of breastfeeding while on PrEP through 6 months
  Proportion of breastfeeding patients with record-reported use of PrEP (oral) at 6-month visit consistent with PrEP metabolite levels consistent with >=4 pills per week among all breastfeeding patients consented to provide samples with record-reported use of PrEP (oral) at 6-month visit and metabolite levels tested

SECONDARY OUTCOMES:
Oral PrEP persistence: Proportion of patients on oral PrEP for 6 months after initiation with no lapse of PrEP coverage exceeding 14 days | PrEP initiation or initiation of breastfeeding while on PrEP through 6 months
  Proportion of breastfeeding patients with health record-reported oral PrEP use who maintain ongoing PrEP usage with no more than a 14-day lapse of expected available pills from oral PrEP approximately 6 months after PrEP initiation, among the total number of breastfeeding patients with health record-reported oral PrEP use
Injectable PrEP persistence: Proportion of patients on injectable PrEP for 6 months after initiation with no lapse of PrEP coverage exceeding 14 days | PrEP initiation or initiation of breastfeeding while on PrEP through 6 months
  Proportion of breastfeeding patients with health record-reported injectable PrEP use who maintain ongoing PrEP usage with no more than a 14-day lapse of timely injections from injectable PrEP approximately 6 months after PrEP initiation, among the total number of breastfeeding patients with health record-reported injectable PrEP use
PrEP persistence: Proportion of patients on PrEP for 12 months after initiation with no lapse of PrEP coverage exceeding 14 days | PrEP initiation or initiation of breastfeeding while on PrEP through 12 months
  Proportion of breastfeeding patients with health record-reported PrEP use (oral or injectable) who maintain ongoing PrEP usage with no more than a 14-day lapse from oral or injectable PrEP at 12 months, among the total number of breastfeeding patients with health record-reported PrEP use (oral or injectable)
Oral PrEP adherence: Proportion of patients on oral PrEP with PrEP metabolite levels consistent with >=4 pills per week at a 12-month oral PrEP visit | PrEP initiation or initiation of breastfeeding while on PrEP through 12 months
  Proportion of breastfeeding patients with record-reported use of PrEP (oral) at 12-month visit with PrEP metabolite levels consistent with >=4 pills per week among all breastfeeding patients consented to provide samples with record-reported use of PrEP (oral) at 12-month visit and metabolite levels tested
Adoption: Number of referrals from all sources to CFL peer mothers | From study start through study end (approximately 3.5 years)
  Number of referrals to CFL peer moms based on CFL peer mom tracking systems across all intervention sites assessed via repeat cross-sectional surveys from study start to study end
Adoption: Number of referrals from PrEP providers to CFL peer mothers | From study start through study end (approximately 3.5 years)
  Number of referrals from PrEP providers to CFL peer mothers based on CFL peer mother tracking systems across all intervention sites assessed via repeat cross-sectional surveys from study start to study end

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Rutstein, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Project Malawi (UNCPM), Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina (UNC).
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Rutstein SE, Lucas VA, Hosseinipour MC, Herce ME, Edwards J, Cassidy C, Villiera J, Kamanga F, Chagomerana M, van Oosterhout JJ, Chikuse E, Rambiki E, Thawani A, Malewezi B, Makhupula L, Udedi C, Mbulaje P, Matoga M, Kumwenda W, Mvalo T, Bula A, Nkhalamba L, Mofolo I, Chinula L, Thonyiwa V, Kumwenda O, Chisema MN, Hoffman IF, Miller WC, Go VF, Pence B, Squibb MA, Saidi F. Leveraging infant visit PrEP screening INtegration & tasK shifting to improve post-partum HIV prevention in Malawi (LINK): a cluster-randomized trial evaluation of a postpartum HIV prevention package among breastfeeding women in Malawi. BMC Health Serv Res. 2025 Aug 19;25(1):1107. doi: 10.1186/s12913-025-13133-6. PMID 40830473